CLINICAL TRIAL: NCT04809129
Title: Testing the Gravitostat in Humans: the Impact of a Weighted Vest in Patients Post Bariatric Surgery on Fat-free Mass Retention and Weight Loss
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding stopped.
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS20-012
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: Bariatric surgery; Obesity; Weight loss maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External mechanical loading (Experimental): Following bariatric surgery (RYGB or SG) patients will be asked to wear a weighted vest for a minimum of 8 hours daily and during physical exercise for three months postoperatively.
  Weight will be incrementally added on a weekly basis to maintain the baseline weight as patients lose weight following surgery up to a maximum of 15%.
  Interventions: Device: Weighted vest
- Standard postoperative care (No Intervention): Patients following bariatric surgery (RYGB or SG) will receive standard postoperative care.

INTERVENTIONS:
Device: Weighted vest — Patients will wear a weighted vest following bariatric surgery with weight increased incrementally to maintain baseline weight. This vest will be worn for a minimum of 8 hours a day for three months postoperatively.
  Arms: External mechanical loading

SUMMARY:
The mechanisms regulating fat mass homeostasis are incompletely understood although recent animal and human trials would suggest that there is a leptin independent regulatory pathway which may play a role in weight control and maintenance. Although evidence would suggest that external loading in patients with obesity may promote body weight loss, this has not been explored in patients following bariatric surgery.

The aim of this study is to investigate the mechanisms regulating weight loss and the potential role of the 'gravitostat' in fat free mass retention in patients following bariatric surgery.

DETAILED DESCRIPTION:
The aim of the study is to investigate the mechanisms that regulate weight loss, particularly following bariatric surgery. Previous animal studies have suggested that there is an underlying regulatory process controlled by 'the gravitostat' which is an evolutionary adaptation responsible for weight control and maintenance. Studies exploring this concept in rodent models have suggested that artificially increasing the animal's weight with the implantation of weighted capsules results in greater weight loss in mice with obesity but does not affect those of normal weight. We will use weighted vests in patients following surgery to replicate this increased mechanical loading to determine whether a similar process occurs in humans. This will improve our understanding of the underlying processes regulating weight in patients with obesity and following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing bariatric surgery- Roux en Y gastric bypass or sleeve gastrectomy
* Age 18-60
* BMI >30kg/m2
* Reporting regular physical exercise (>3 days/week)
* Willingness to comply with the study protocol

Exclusion Criteria:

* Sedentary lifestyle
* Chronic pain that is constant and impairs the quality of life such as severe back, hip or knee pain
* Reduced mobility requiring the use of a mobility aid
* Undergoing revisional surgery
* Concerns from the investigator that the participant will be unable to fully comply with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-10-03 (Estimated); Study Completion 2022-10-03 (Estimated)

PRIMARY OUTCOMES:
Fat free mass retention | 1 year
  Fat free mass retention as measured using DEXA scan
Weight loss | 1 year
  Weight loss (kg)

SECONDARY OUTCOMES:
Changes in protein and inflammatory marker levels myostatin | 1 year
  Change in myostatin
Changes in protein and inflammatory markers lipocalin-2 | 1 year
  Change in lipocalin-2
Changes in protein and inflammatory markers IGF-1 | 1 year
  Change in IGF-1
Changes in protein and inflammatory markers IL-6 | 1 year
  Change in IL-6
Changes in protein and inflammatory markers | 1 year
  Change in testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Carel W le Roux, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin Clinical Research Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No